CLINICAL TRIAL: NCT05564663
Title: Testing a PTSD m-Health Intervention to Improve Alcohol Treatment Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kipling Bohnert, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00006258; R01AA028213 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD Coach App + Brief Support (Experimental): PTSD Coach App + Brief Support will include brief instruction and support for the use of the PTSD Coach App developed by the study team. The PTSD Coach App incorporates evidence-based assessment, psychoeducation, and self-management strategies for PTSD symptoms that are customizable to the user.
  Interventions: Behavioral: PTSD Coach App + Brief Support
- Enhanced Usual Care (EUC) (Active Comparator): EUC will include brief psychoeducation regarding PTSD and alcohol use disorder (AUD) and resources for PTSD-related mental health treatment.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: PTSD Coach App + Brief Support — PTSD Coach App + Brief Support will include downloading the PTSD Coach App for personal use and four, brief (<20 minutes), weekly, individual support sessions. The sessions will focus on the instruction and encouragement of App use and activities (i.e., assessments, self-management strategies, and psychoeducational readings).
  Arms: PTSD Coach App + Brief Support
Behavioral: Enhanced Usual Care (EUC) — EUC will consist of one brief session (with brochure) of PTSD and AUD psychoeducation and referral information for mental health clinics that provide PTSD services, with encouragement to schedule an appointment at one of the listed clinics to discuss PTSD-related symptoms.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The purpose of this study is to learn whether a mobile health application (mHealth App) for posttraumatic stress disorder (PTSD) with brief support can help individuals who are in treatment for alcohol problems.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Currently in addictions treatment
* Meet criteria for a current Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) AUD diagnosis
* A score of 33 or greater on the PTSD Checklist (PCL-5)
* Own a smart phone or other type of Wi-Fi-enabled device with App capabilities

Exclusion Criteria:

* Injection drug use in the past year
* Patients who are unable to speak and/or understand English
* Patients who are currently engaged in specific therapy for PTSD (Prolonged Exposure Therapy, Cognitive Reprocessing Therapy, EMDR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) Change | Baseline, 1-, 3-, 6-, and 12-months
  The PCL-5 is a 20-item, self-reported measure that assesses the 20 DSM-5 symptoms of PTSD. Each symptom is measured on a 0-4 scale, with higher values indicating greater severity. Total scale scores range from 0 to 80.
Timeline Followback (TLFB) for Alcohol Change | Baseline, 1-, 3-, 6-, and 12-months
  The TLFB assessment method will be used to assess alcohol use in the past 30-days.

CONTACTS AND LOCATIONS:
Overall Officials: Kipling Bohnert, Principal Investigator — Michigan State University
Locations (1):
- Pine Rest Christian Mental Health Services, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No